CLINICAL TRIAL: NCT06661291
Title: Utilization of Digital Health Platform Plus Live Coaching Improves Surgical Patients Outcomes - Phase II
Brief Title: Pip Care to Improve Surgical Patient Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jennifer Holder-Murray, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY25010036; R42HL174371 (NIH)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Abdominal Surgery

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial to determine the effectiveness of Pip Care in improving clinical and patient reported outcomes when compared to standard perioperative care in 1300 subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pip Care Intervention Group (Experimental): Subjects randomized to the Pip Care Intervention group will receive access to the Pip Care digital health platform 1-week prior to their scheduled elective, inpatient surgery and retain access to the digital health platform for 30-days following surgery.
  Interventions: Other: Pip Care Digital Health Platform
- Standard of Care Group (Active Comparator): Subjects randomized to the standard of care group will receive routine standard of care for their planned elective, inpatient surgery.
  Interventions: Other: Standard of Care Protocol

INTERVENTIONS:
Other: Pip Care Digital Health Platform — Pip Care Digital Health Platform is a smartphone application granting access to a health coach who will assist the patient in completing a health intake, creating personalized perioperative care plans, and meets regularly with the patient to encourage goal accomplishments and supports healthy surgical recovery.
  Arms: Pip Care Intervention Group
Other: Standard of Care Protocol — Subjects in this intervention group will receive routine, standard of care throughout their surgery and hospital stay as determined by their acting clinical care team.
  Arms: Standard of Care Group

SUMMARY:
Pip Care is developing a personalized, interactive surgical journey platform with a live health coach that works directly with health systems to optimize the perioperative care process. Our Health Insurance Portability and Accountability Act (HIPAA)-compliant platform, Pip, can be integrated into any electronic medical record (EMR), thus alleviating the administrative burden by making operational workflows more efficient. The PIP empowers patients and their families to be more involved in their care by breaking down a patient's healthcare plan into definable, easy-to-understand, and easy-to-complete tasks. Additionally, a health coach completes a health intake to create a personalized perioperative care plan, meets regularly with the patient to encourage goal accomplishment, and facilitates care coordination. This project has 2 phases; Phase I is to assess usability of the Pip Care platform in surgical patients, Phase II is a RCT (Randomized Controlled Trial) to assess surgical clinical outcomes while using Pip compared to standard of care.

DETAILED DESCRIPTION:
In the United States (US), 48 million surgeries are performed annually, and despite medical and surgical advancements, postoperative complications are the third leading cause of death. Perioperative risk varies between patients based on their health and surgical procedure. Patients with intermediate or high perioperative risk experience extended hospital stays, higher readmission rates, and frequent adverse events, including death. The national burden for such cases costs $31.35 billion annually. As a result, the healthcare industry is prioritizing the advancement of perioperative care to reduce postoperative complications and improve patient outcomes. While clinical care teams provide clinical pathways for patients, patients find the perioperative journey complex and impersonal. Patients often don't have access to a tailored preparation plan and personal guidance, emotional support, and motivation despite the high level of perioperative care detail and the vulnerable status of patients. Therefore, there is an unmet need to provide patients with comprehensive perioperative care guidance and support with the enhanced human touch to reduce postoperative complications. Integrating clinical pathways prepared by interdisciplinary care teams and digital health platform offers opportunities to improve patient outcomes through improved prehabilitation and postoperative engagement.

PRELIMINARY DATA:

The first version of Pip included three pathways (nutrition, fitness, and smoking cessation). In a pilot study with the Center for Perioperative Center (CPC) at the University of Pittsburgh Medical Center (UPMC), implementation of Pip resulted in the reduction of the median length of stay (LOS) by one day. The same-day surgery cancellations were avoided 99.5 % of the time. Pip also received an aggregate patient satisfaction score of 4.8 out of 5 (vs. industry benchmarks of 3.8-4.3).

Pip Care partnered with the UPMC CPC to digitize and implement clinical pathways, created by perioperative experts at UPMC, into modular digital care contents. Pip Care, CPC, and surgical offices developed a workflow that was both operationally and clinically seamless. The Pip DHP was designed to replace the time-consuming clinic follow-ups and care coordination through the different phases of the perioperative process. In addition to Health Coach follow-up, patients were invited to not only receive notifications and report outcomes, but to explore a library of educational multimedia resources on disease processes and why optimization of said diseases is important prior to surgery. Pip also identified patients who were not engaging with the clinical team and offered further remediation to help prevent poor outcomes.

Pip Digital Platform Development. The Pip technology platform is powered by two connected components: (1) Back-end platform utilized by health coaches and (2) Front-end native digital mobile application utilized by patients. The front-end digital mobile application contains four key features, which are represented by separate pages within the digital application: (1) Pip My Plan, which displays when patients are assigned personalized care plans and tasks by their Health Coach, (2) Pip Appointments, which patients schedule and join weekly video or voice calls with the Health Coach, (3) Pip Messages patients have access to unlimited engagement with their Health Coach, and (4) a library of health system-approved education content, including articles and videos, to assist with their surgery preparation and recovery. Figure 4 summarizes the initial Pip care plans: 8 total care plans including 3 clinical pathways (smoking cessation, weight management, and nutrition). To make the application patient-centered and accessible to all with mobile technology while improving communication, language for the application (e.g., questions, answers, instructions), and other content within the application are presented at a maximum reading level of the eighth grade. Pip is designed to function on both iOS (Apple Inc, Cupertino, CA) and Android (Google Inc, Mountain View, CA) operating systems.

Case Matched Pilot Clinical Study. A pilot clinical study at UPMC recently demonstrated feasibility and improved outcomes in case matched patients. The investigators have developed and validated the feasibility of the Pip Care digital platform with Health Coach and digital protocols. This was a Quality Improvement approved descriptive, prospective feasibility study of patients scheduled for elective surgery, invited to enroll in Pip from 2.5-4 weeks preoperatively through 4 weeks postoperatively at UPMC between 11/2/2022 - 3/27/2023. Descriptive primary endpoints included patient satisfaction, patient engagement, Pip Health Coach evaluations, and other PROs. Secondary endpoints included length of stay (LOS), readmission rates, and emergency department utilization rates within 30 days. Mean age was 64 years.

High Engagement and Satisfaction Scores. Our primary outcomes focused on feasibility of deployment of the combined platform and the patient assessment of the experience. Out of 283 patients invited to Pip, 172 patients (61%) were enrolled compared to industry benchmarks between (5% and 30%). Of those enrolled, 143 (83%) had one or more Health Coach sessions. During the study, of the patients who had one or more Health Coach sessions, 138 (97%) proceeded to surgery, a 4-8% improvement compared to industry benchmarks (90-93%). After surgery, 97 (70%) patients engaged with Pip postoperatively, a 35-126% improvement compared to industry benchmarks (31-52%). Pip received a total of 95 patient satisfaction survey submissions. Patients reported an overall high satisfaction based on the satisfaction survey (average score 4.8 out of 5, n=95). Patients strongly agree that Health Coach helped them throughout the perioperative process based on Pip Health Coach evaluation (average score 4.97 out of 5, n=33). The average Net Promotor Score, a customer experience metric, was 9.7 out of 10.

LOS and Readmission. Stabilized inverse probability of treatment weighting (SIPTW) was created to reduce selection bias and balance the patient characteristics (i.e., age, procedures, and perioperative risk score) in Pip and non-Pip cohorts. A total of 128 patients in the Pip cohort were compared to 268 patients in the non-Pip cohort. Pip was significantly associated with a 24% reduction in postoperative LOS (mean 2.4 vs. 3.1 days; median 1.9 vs. 3.0 days; mean ratio: 0.76; 95%CI: 0.62-0.93). Pip was associated with a 49% lower risk in 7-day readmission (relative risk: 0.51; 95%CI: 0.11-2.31) and 17% lower risk in 30-day readmission (relative risk: 0.83; 95%CI: 0.30-2.31), though not statistically significant. Pip and non-Pip groups had similar risk in 30-day ED returns (relative risk: 1.06; 95%CI: 0.56-2.01).

Patient Feedback to the Health Coach. An overwhelmingly positive aspect was the patient feedback and response to the Health Coach. The following comments support current evidence that high level engagement is very important to patients and their outcomes

"This has been a medical experience I will not forget. [The Health Coach] was patient and kind and encouraging. His support was vital to my experience." - Patient

"Talking to [the Health Coach] has helped me to feel a bit better and know that I am doing all that is in control to get ready for surgery." - Patient

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient ≥18 years old
2. Planned elective, inpatient surgery between 2 to 8 weeks following enrollment in Pip within the following surgical specialties: complex abdominal surgery (general surgery, colorectal surgery, surgical oncology), gynecologic oncology, thoracic surgery, spine surgery, and orthopedic joint surgery
3. Daily access to a smartphone or tablet.

Exclusion Criteria:

1. Unable to speak English
2. Unable to use a smartphone or tablet independently or with daily assistance.
3. Currently pregnant (assessed via standard-of-care pre-operative workup)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay | Up to 7 days following surgery
  The total length of hospital stay (# of days) compared between study groups. Outcome will be reported as mean(SD).
Hospital Readmission | Up to 30 days following surgery
  This outcome will be measured by the count of participants who experience hospital readmission following surgery in each study group.

SECONDARY OUTCOMES:
Emergency Room Visits Post-Operatively | Up to 30 days following surgery
  This outcome will be measured by % of participants per group who have visited the emergency room following hospital discharge in their 30-day study participation.
Discharge to Long-term Care Facility | Up to 30 days following surgery
  This outcome will be measured by % of participants per group who have been discharged to a long-term care facility following hospital discharge in their 30-day study participation.
Complication Rates | Up to 30 days following surgery
  This outcome will be measured by the count of participants per group who have experienced any surgery-related complications during their 30-day study participation. Complication experiences will be tracked by yes - subject has experienced one or more complications, or no - subject has not experienced any complications.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Holder-Murray, MD, Principal Investigator — University of Pittsburgh, UPMC
Locations (8):
- United States (8):
  - UPMC Jameson Hospital, New Castle, Pennsylvania
  - UPMC East Hospital, Pittsburgh, Pennsylvania
  - UPMC Horizon, Pittsburgh, Pennsylvania
  - UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Passavant Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with others inside and outside of the University who are conducting similar research. Though, at this time, there is no plan to share data with outside universities.
  De-identified data will be shared with PIP CARE INC.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available as soon as it is retrieved per subject and will be available for 3.5 years (duration of the study enrollment and one year after for data analysis purposes)
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).